CLINICAL TRIAL: NCT05339620
Title: Effect of Implant Driver Facilitated Micro-osteo Perforations on the Rate of Tooth Movement.
Brief Title: Effect of Implant Driver Facilitated Micro-osteo Perforation on the Rate of Tooth Movement.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahria University (Other)
Responsible Party: Principal Investigator, DR MARIA HABIB, Assistant Professor, Bahria University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ERC 05/2018
Record Dates: First submitted 2022-04-15; First posted 2022-04-21 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Tooth Movement Techniques
Keywords: micro-osteoperforations, tooth movement, implant driver

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mop group (Experimental): a group of patients with a class 2 divsion 1 dental malocclusion, overjet greater than 9 mm, extraction of upper first premolars planned, and it has been 3 months post extraction and before canine retraction is commenced.
  Interventions: Procedure: implant driver facilitated micro-osteoperforations
- mop group ( same) (Active Comparator): a group of patients with a class 2 divsion 1 dental malocclusion, overjet greater than 9 mm, extraction of upper first premolars planned, and it has been 3 months post extraction and before canine retraction is commenced.
  Interventions: Procedure: implant driver facilitated micro-osteoperforations

INTERVENTIONS:
Procedure: implant driver facilitated micro-osteoperforations — 3 micro-osteoperforations(in a vertical pattern) are done on the randomly allocated experimental side , distal to canine under local anesthesia. the other side of the mouth is used as a control.
  alginate impression is taken before the intervention .
  Other Names: micro-osteoperforations by any other means.

SUMMARY:
we have conducted a split-mouth randomized clinical trial to study effects of implant induced micro-osteoperforations on the rate of tooth movement during canine retraction.

DETAILED DESCRIPTION:
The experimental group will receive implant driver facilitated microosteoperforation on one side of the mouth( according to split mouth design) decided by random allocation.

After 3 months of extraction of upper first premolar ( according to planned orthodontic treatment), 3 microosteoperforation will be done with implant in an implant driver distal to canine. Surgical procedure will be done in local anesthesia, no flap will be raised. Alginate impressions will be taken before the procedure and 28 days after canine retraction has started, to measure the difference between rate of canine retraction on both sides. Measurement was done by a digital vernier caliper,

ELIGIBILITY:
Inclusion Criteria:

* • Male and female

  * Age 18- 45 years
  * Class 2 div 1
  * No systemic disease
  * No radiographic evidence of bone loss
  * No history of periodontal therapy
  * No current active periodontal disease
  * No smoking
  * No gingivitis or untreated caries
  * Probing depth < 4mm in all teeth
  * Gingival index < 1mm
  * Plaque index < 1mm

Exclusion Criteria:

* Long term use of antibiotics, phenytoin,cyclosporine, anti inflammatory drugs, systemic corticosteroids and calcium channel blockers.
* Poor oral hygiene for more than 2 visits.
* Extreme skeletal class 2 malocclusion, overjet > 10mm, anb> 7
* Systemic disease
* Evidence of bone loss
* Past periodontal disease
* Current periodontal disease
* Smoking
* Gingivitis and caries
* Probing depth > 4mm

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2018-01-07 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-03-20 (Actual)

PRIMARY OUTCOMES:
Comparing rate of canine retraction between intervention and non-intervention side. | 28 days
  distance from cusp tip of canine to mesio-buccal cusp tip of molar taken by digital vernier caliper.

CONTACTS AND LOCATIONS:
Locations (1):
- Bahria University Medical and Dental College, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cheung T, Park J, Lee D, Kim C, Olson J, Javadi S, Lawson G, McCabe J, Moon W, Ting K, Hong C. Ability of mini-implant-facilitated micro-osteoperforations to accelerate tooth movement in rats. Am J Orthod Dentofacial Orthop. 2016 Dec;150(6):958-967. doi: 10.1016/j.ajodo.2016.04.030. PMID 27894545
- [Background] Ozkan TH, Arici S. The effect of different micro-osteoperforation depths on the rate of orthodontic tooth movement: A single-center, single-blind, randomized clinical trial. Korean J Orthod. 2021 May 25;51(3):157-165. doi: 10.4041/kjod.2021.51.3.157. PMID 33984223
- [Background] Aboalnaga AA, Salah Fayed MM, El-Ashmawi NA, Soliman SA. Effect of micro-osteoperforation on the rate of canine retraction: a split-mouth randomized controlled trial. Prog Orthod. 2019 Jun 3;20(1):21. doi: 10.1186/s40510-019-0274-0. PMID 31155698
- [Background] Bolat Gumus E, Kinsiz E. Effects of miniscrew-facilitated micro-osteoperforations on the rate of orthodontic tooth movement : A split-mouth, randomized controlled trial. J Orofac Orthop. 2023 Apr;84(Suppl 2):104-110. doi: 10.1007/s00056-021-00371-6. Epub 2022 Jan 13. PMID 35024875